CLINICAL TRIAL: NCT03570424
Title: Whey Protein Support to Metabolic and Performance Adaptations in Response to High Intensity Interval Training in Young Adult Men
Brief Title: Whey Protein Support to Metabolic and Performance Adaptations in Response HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Brian Carson, Lecturer in Exercise Physiology, University of Limerick, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7867835
Record Dates: First submitted 2018-05-22; First posted 2018-06-27 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Muscle, Skeletal; High-Intensity Interval Training; Exercise
Keywords: Organelle Biogenesis; Adaptation, Physiological; Whey Proteins; Protein Hydrolysates
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomly assigned, parallel group, simple pre-post design has been adopted to answer this question. 3 groups of young (aged 18-35 y), healthy, recreationally active, aerobically untrained (VO2max <50 ml.kg.min-1) males will undertake 3 weeks (9 sessions) of HIIT under different nutrient conditions following >10h overnight fast: i) Fasted placebo (0.33g.kg-1 body artificially flavoured and textured placebo); ii) Fed Whey protein (0.33g.kg-1 body mass intact whey protein 45 minutes prior to exercise); iii) Fed Whey protein hydrolysate (0.33g.kg-1 body mass hydrolysed whey protein 45 minutes prior to exercise). Participants will undergo biological sampling (venous blood and muscle biopsy) and measures of performance pre and post the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are block randomised to one of three nutrient conditions on provision of informed consent. This information is held by the PI and members of the research team independent of the outcomes assessor (masked). All three beverages are made up by members of the research team independent of the outcomes assessor (masked) and the participants (masked). Each participant (masked) is provided with a drink in a black, non-transparent, container with no details of its contents other than that is a "nutrient supplement".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Intervention (Nutrient support to HIIT): Participants consume 0.33g.kg-1 body mass of artificially flavoured and textured placebo 45 minutes prior to HIIT exercise
  Interventions: Dietary Supplement: Placebo
- Whey Protein (Experimental): Intervention (Nutrient support to HIIT): Participants consume 0.33g.kg-1 body mass intact whey protein 45 minutes prior to HIIT exercise
  Interventions: Dietary Supplement: Nutrient support to HIIT
- Whey Protein Hydrolysate (Experimental): Intervention (Nutrient support to HIIT): Participants consume 0.33g.kg-1 body mass hydrolysed whey protein 45 minutes prior to HIIT exercise
  Interventions: Dietary Supplement: Nutrient support to HIIT

INTERVENTIONS:
Dietary Supplement: Nutrient support to HIIT — 3 groups of young (aged 18-35 y), healthy, recreationally active, aerobically untrained (VO2max <50 ml.kg.min-1) males will undertake 3 weeks (9 sessions) of HIIT under different nutrient conditions following >10h overnight fast: i) Placebo: Fasted artificially flavoured and textured placebo 45 minutes prior to exercise; ii) Whey protein 45 minutes prior to exercise; iii) Whey protein hydrolysate 45 minutes prior to exercise).
  Arms: Whey Protein; Whey Protein Hydrolysate
Dietary Supplement: Placebo — 3 groups of young (aged 18-35 y), healthy, recreationally active, aerobically untrained (VO2max <50 ml.kg.min-1) males will undertake 3 weeks (9 sessions) of HIIT under different nutrient conditions following >10h overnight fast: i) Fasted artificially flavoured and textured placebo 45 minutes prior to exercise; ii) Fed Whey protein 45 minutes prior to exercise; iii) Fed Whey protein hydrolysate 45 minutes prior to exercise).
  Arms: Placebo

SUMMARY:
High intensity interval training (HIIT) has recently emerged as a time efficient alternative to conventional endurance exercise, conferring similar or superior benefits in terms of metabolic and performance adaptations in both athletic and non-athletic populations. Some of these physiological adaptations include augmented mitochondrial biogenesis and improved substrate metabolism in peripheral tissues such as skeletal muscle. However, nutritional strategies to optimise the adaptations to HIIT have yet to be established. Recent evidence suggests that acute nutritional status can affect the molecular regulation of genes mediating substrate metabolism and mitochondrial biogenesis. Moreover, preliminary evidence suggests that completion of exercise in fasted conditions augments some of these exercise-induced adaptations compared with the fed state. Given the fact that the transient molecular adaptations to acute exercise mediate long-term physiological adaptations, an investigation into the effects of different nutritional interventions on metabolic and performance responses to HIIT is warranted.

The purpose of this study is to determine the effects of fasted vs. fed-state (Whey Protein) HIIT on metabolic and performance adaptations in the acute (single exercise session) and chronic (3 weeks, 9 exercise sessions) phases. The primary hypothesis is that different pre-exercise feeding conditions (e.g. fasted placebo vs. Whey protein fed) will result in divergent physiological adaptations in terms of skeletal muscle metabolism and performance, both in response to a single HIIT session and a chronic HIIT intervention.

DETAILED DESCRIPTION:
High intensity interval training (HIIT) has recently emerged as a time efficient alternative to conventional endurance exercise, conferring similar or superior benefits in terms of metabolic and performance adaptations in both athletic and non-athletic populations. Some of these physiological adaptations include augmented mitochondrial biogenesis and improved substrate metabolism in peripheral tissues such as skeletal muscle. However, nutritional strategies to optimise the adaptations to HIIT have yet to be established. Recent evidence suggests that acute nutritional status can affect the molecular regulation of genes mediating substrate metabolism and mitochondrial biogenesis. Moreover, preliminary evidence suggests that completion of exercise in fasted conditions augments some of these exercise-induced adaptations compared with the fed state. Given the fact that the transient molecular adaptations to acute exercise mediate long-term physiological adaptations, an investigation into the effects of different nutritional interventions on metabolic and performance responses to HIIT is warranted.

The purpose of this study is to determine the effects of fasted vs. fed-state (Whey Protein) HIIT on metabolic and performance adaptations in the acute (single exercise session) and chronic (3 weeks, 9 exercise sessions) phases. The primary hypothesis is that different pre-exercise feeding conditions (e.g. fasted vs. Whey protein fed) will result in divergent physiological adaptations in terms of skeletal muscle metabolism and performance, both in response to a single HIIT session and a chronic HIIT intervention.

A randomly assigned, parallel group, simple pre-post design has been adopted to answer this question. 3 groups of young (aged 18-35 y), healthy, recreationally active, aerobically untrained (VO2max <50 ml.kg.min-1), protein sufficient (>0.8 g.kg.d-1), males will undertake 3 weeks (9 sessions) of HIIT under different nutrient conditions following >10h overnight fast: i) Fasted placebo (0.33g.kg-1 body mass artificially flavoured and textured placebo); ii) Fed Whey protein (0.33g.kg-1 body mass intact whey protein 45 minutes prior to exercise); iii) Fed Whey protein hydrolysate (0.33g.kg-1 body mass hydrolysed whey protein 45 minutes prior to exercise). Participants will undergo biological sampling (venous blood and muscle biopsy) and measures of performance pre and post the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (absence of clinical condition)
* Recreationally active
* Aerobically untrained (VO2max <50 ml.kg.min-1)
* Protein sufficient (>0.8 g.kg.d-1)
* Males
* Able to provide informed consent
* No contraindications to high intensity exercise

Exclusion Criteria:

* BMI >30 kg.m-2
* Metabolic disease (mitochondrial, Type 2 Diabetes)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Organelle Biogenesis (Mitochondrial) Acute | Acute - 3 hours post exercise session 1
  Acute phase - change in Peroxisome Proliferator Activated Receptor 1 alpha (PGC-1α) messenger ribonucleic acid (mRNA) expression in response to a single HIIT session. Measured using real-time polymerase chain reaction (RT-PCR).
Exercise Performance | Chronic - 72 hours post exercise session 9
  Mean power output (Watts) during 20 minute cycling performance test. Measured using cycle ergometer and associated software.
Anaerobic Exercise Performance | Chronic - 72 hours post exercise session 9
  Anaerobic exercise performance peak power (Watts). Measured using 30 second Wingate test on a Monark 894E cycle ergometer.
Organelle Biogenesis (Mitochondrial) Chronic | Chronic - 48 hours post exercise session 9
  Chronic Phase - change in Citrate Synthase Activity measured using commercially available assay kits.

SECONDARY OUTCOMES:
Organelle Biogenesis (Mitochondrial) | Acute: 3 hours post HIIT session 1.
  Pyruvate Dehydrogenase Kinase 4 (PDK4), Peroxisome Proliferator Activated Receptor (PPAR) delta, Sirtuin 1 (SIRT1) mRNA expression. Measured using real-time polymerase chain reaction (RT-PCR).
Cycling Economy | Chronic - 72 hours post exercise session 9
  Cycling economy (W.VO2 L.min-1) during multiple incremental stages (50 W, 100 W, 150 W, 200 W, 250 W) of a submaximal cycling test.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Carson, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03570424/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03570424/ICF_002.pdf